CLINICAL TRIAL: NCT03864406
Title: Impact of Steady State Cobicistat and Darunavir/Cobicistat on the Pharmacokinetics and Pharmacodynamics of Oral Anticoagulants (Rivaroxaban, Apixaban) in Healthy Volunteers
Brief Title: Impact of Steady State Cobicistat and Darunavir/Cobicistat on the Pharmacokinetics and Pharmacodynamics of Oral Anticoagulants (Rivaroxaban, Apixaban) in Health Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 190063; 19-CC-0063
Record Dates: First submitted 2019-03-05; First posted 2019-03-06 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers
Keywords: Antiretroviral Therapy; Human Immunodeficiency Disease; Drug-Drug Interactions; Thrombosis; Bleeding
MeSH Terms: conditions — Thrombosis; Hemorrhage | interventions — Cobicistat; cobicistat mixture with darunavir; Rivaroxaban

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pharmacokinetic study in healthy volunteers (Experimental): Healthy participants received a single dose of rivaroxaban 10 mg orally on day 1 (phase 1) followed by cobicistat 150 mg once daily from days 2 - 7 and a single dose of rivaroxaban 10 mg on day 7 (phase 2). Participants received darunavir /cobicistat 800/150 mg once daily from days 8 - 13 followed by a single dose of rivaroxaban 10mg on day 13 (phase 3). Serial blood sampling was done on days 1, 7, and 13.
  Interventions: Drug: Cobicistat; Drug: Darunavir/Cobicistat; Drug: Rivaroxaban

INTERVENTIONS:
Drug: Cobicistat — Each tablet of Tybost contains 150 mg of cobicistat.
  Other Names: Tybost
Drug: Darunavir/Cobicistat — Each tablet of Prezcobix contains 800 mg of darunavir and 150 mg of cobicistat.
  Other Names: Prezcobix
Drug: Rivaroxaban — Each tablet of Xarelto contains 10 mg of rivaroxaban.
  Other Names: Xarelto

SUMMARY:
Background:

Rivaroxaban and apixaban are blood thinners. People with HIV may need to take them to treat or prevent blood clots. The anti-HIV drug darunavir (DRV) can increase the amount of these blood thinners in the body. This can cause bleeding or other health problems. The drug cobicistat (COBI) is used to help anti-HIV drugs work better. Researchers want to give healthy people DRV combined with COBI to learn how it affects rivaroxaban or apixaban blood levels.

Objective:

To test blood levels of rivaroxaban or apixaban when taken with COBI and DRV/COBI.

Eligibility:

Healthy volunteers ages 18-65

Design:

Participants will be screened with:

Medical history

Physical exam

Fasting blood and urine tests. (Urine tests will be performed in females of child-bearing potential only)

Participants will have 8 visits; 3 are long (about 10-12 hours) and 5 are about 1 hour. They include:

Baseline and final visits:

Fasting blood and urine tests

Day 1 visit (long day):

Fasting blood and urine tests

Catheter placement: A needle will insert a small tube into the participant's arm vein. Blood will be drawn up to 10 times.

Dose of rivaroxaban or apixaban

Day 2 visit (short day):

Fasting blood tests

Dose of COBI

Participants will receive a bottle containing COBI tablets to take at home.

Day 7 (long day):

Fasting blood and urine tests

Catheter placement: A needle will insert a small tube into the participant's arm vein. Blood will be drawn up to 10 times.

Dose of rivaroxaban or apixaban

Dose of COBI

Day 8 (short day):

Fasting blood tests

Dose of DRV/COBI Participants will receive a bottle containing DRV/COBI tablets to take at home.

Day 13 (long day):

Fasting blood and urine tests

Catheter placement: A needle will insert a small tube into the participant s arm vein. Blood will be drawn up to 10 times.

Dose of rivaroxaban or apixaban

Dose of DRV/COBI

Day 14 (short day):

Fasting blood tests

Participants will take COBI tablets daily at home on days 3-6, and DRV/COBI on days 9 -12 during the study. They will record doses and side effects.

During the study, participants cannot:

Take most medications.

Drink alcohol, smoke, or vape

Engage in activities such as contact and extreme sports

DETAILED DESCRIPTION:
Rivaroxaban is a direct oral anticoagulant (DOAC) used for the prevention and treatment of various thromboembolic disorders. Predictable pharmacokinetic (PK) and pharmacodynamic (PD) properties, coupled with a few drug drug and food-drug interactions, distinguishes DOACs from a traditionally used anticoagulant, warfarin, allowing fixed dosing without routine coagulation monitoring. Patients with human immunodeficiency virus (HIV) are living as long as their HIV negative counterparts due to safe and efficacious antiretroviral therapy (ART). Persons with HIV are at higher risk for thromboembolic events and DOACs are a feasible option for anticoagulation in this population. However, there is a lack of drug interaction and safety data currently on the co-administration cobicistat (COBI)-boosted antiretroviral (ARV) regimens with rivaroxaban. Rivaroxaban is metabolized by cytochrome P450 isozyme (CYP) 3A4 and its absorption is modulated by permeability glycoprotein (P-gp), both of which are inhibited by the PK booster COBI. It is therefore possible that plasma concentrations of rivaroxaban may be significantly increased when co-administered together with COBI. This is of clinical concern as increased anticoagulant exposure may result in bleeding without the security of routine clinical monitoring. The purpose of this study is to determine the effects of steady state concentrations of COBI and darunavir (DRV)/COBI on the PK and PD of single oral doses of rivaroxaban.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject will be considered eligible for this study only if all of the following criteria are met:

* Adults between the ages of 18 to 65 years.
* Body mass index between 18 to 30 kg/M(2).
* Judged to be healthy based on medical history, physical examination, vital signs and clinical laboratory tests (liver function tests (LFTs: alanine transaminase (ALT), aspartate transaminase (AST), total bilirubin less than or equal to upper limit of normal (ULN) (with the exception of participants with Gilbert's syndrome), albumin within normal limits (WNL)], eGFR > 90 mL/min/1.73 m(2), PLT>150,000/microL, hemoglobin (Hgb) greater than or equal to 12 g/dL, activated partial thromboplastin time (aPTT) less than or equal to ULN, partial thromboplastin time (PTT) less than or equal to ULN, international normalized ratio (INR) less than or equal to ULN.
* Subject agrees to storage of specimens for future research.
* Negative serum or urine pregnancy test for females of child-bearing potential.
* For female subjects, willing to avoid pregnancy by (a) practicing abstinence or (b) using effective non-hormonal and/or barrier methods of birth control, as well as avoid breast feeding or providing breast milk to infant during the study period. (baseline visit up to end of study day 20 plus minus 3)
* Willing to avoid engaging in activities such as contact sports, including extreme sports, that may increase the risk of bleeding through body injury or bruising, during the study period (baseline visit up to end of study day 20 plus minus 3)
* Willingness to forgo drinking alcohol during the study period (baseline visit up to end of study day 20 plus minus 3)
* Able to provide consent.

EXCLUSION CRITERIA:

A subject will be ineligible for this study if one, or more, of the following criteria are met:

* HIV infection, as determined by standard serologic or virologic assays for HIV infection.
* Laboratory evidence of active or chronic hepatitis A, B or C infection.
* History or presence of any of the following:

  * any major medical conditions that requires daily frequent medication or potentially impairs medication absorption, metabolism and elimination
  * any other condition that may interfere with the interpretation of the study results, or not be in the best interest of the subject in the opinion of the Investigator.
* Current participation in an ongoing investigational drug protocol or use of any investigational drug within 30 days (based on last dose received) prior to receipt of any study drugs/medications.
* History or presence of the following:

  * bleeding/hematologic disorders (e.g., anemia, hemophilia, etc.),
  * serious/major bleeding event (intracranial, gastrointestinal (GI), as assessed by subject interview), or
  * current increased risk of bleeding
  * for female subjects, menorrhagia
* Planned invasive or surgical procedure within (prior to or following) 28 days of study participation.
* Therapy with any prescription, over-the-counter, herbal, or holistic medications, including hormonal contraceptives by any route, within 5 half-lives of the agent prior to receipt of any study medications will not be permitted with the following exception:

Intermittent or short-course therapy (<14 days) with prescription, vaccines or over-the-counter medications will be reviewed by investigators on a case-by-case basis for potential drug interactions.

* Inability to obtain venous access for sample collection.
* Inability to swallow whole capsules and/or tablets.
* Pregnant female.
* Breastfeeding female.
* The presence of persistent diarrhea or malabsorption that could interfere with the subject's ability to absorb drugs.
* Illicit drug or alcohol use
* Use of nicotine-containing tobacco products, including cigarettes, vaping and chewing tobacco.
* Known hypersensitivity to rivaroxaban, apixaban, COBI or DRV.
* History of documented hypersensitivity to sulfa allergy.
* Organ transplant recipient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen M Hadigan, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not reported or shared. The study team are the only individuals who have access to individual participant data. All data will be analyzed and reported in aggregate.

REFERENCES:
- [Background] Mueck W, Kubitza D, Becka M. Co-administration of rivaroxaban with drugs that share its elimination pathways: pharmacokinetic effects in healthy subjects. Br J Clin Pharmacol. 2013 Sep;76(3):455-66. doi: 10.1111/bcp.12075. PMID 23305158
- [Background] Kumar P, Gordon LA, Brooks KM, George JM, Kellogg A, McManus M, Alfaro RM, Nghiem K, Lozier J, Hadigan C, Penzak SR. Differential Influence of the Antiretroviral Pharmacokinetic Enhancers Ritonavir and Cobicistat on Intestinal P-Glycoprotein Transport and the Pharmacokinetic/Pharmacodynamic Disposition of Dabigatran. Antimicrob Agents Chemother. 2017 Oct 24;61(11):e01201-17. doi: 10.1128/AAC.01201-17. Print 2017 Nov. PMID 28848011
- [Background] Frost C, Nepal S, Wang J, Schuster A, Byon W, Boyd RA, Yu Z, Shenker A, Barrett YC, Mosqueda-Garcia R, Lacreta F. Safety, pharmacokinetics and pharmacodynamics of multiple oral doses of apixaban, a factor Xa inhibitor, in healthy subjects. Br J Clin Pharmacol. 2013 Nov;76(5):776-86. doi: 10.1111/bcp.12106. PMID 23451769
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-CC-0063.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Versus Time Curve (AUC0-∞) for Rivaroxaban
Description: Area under the concentration versus time curve from 0 to infinity (AUC0-∞) following a single dose of rivaroxaban 10 mg orally on days 1, 7, and 13 to measure the total drug exposure was analyzed by the linear up/log down trapezoidal rule using noncompartmental methods with Phoenix WinNonlin® (version 8.0; Pharsight Corporation, Mountain View, CA).
Time Frame: Total drug exposure at time point zero to infinity on days 1, 7, & 13
Population: All participants who completed at least one intensive pharmacokinetic visit were included in the pharmacokinetics analysis
Measure: Mean (Standard Deviation); unit: hr*ng/ml
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 12
hr*ng/ml
  Day 1 (phase 1) | 1049.19 (401.58)
  Day 7 (phase 2) | 2274.3 (766.51)
  Day 13 (phase 3) | 2226.38 (918.07)

2. Primary Outcome: Area Under the Concentration Versus Time Curve (AUC0-24hr) for Rivaroxaban
Description: Area under the concentration versus time curve from (AUC0-24hr) following a single dose of rivaroxaban 10 mg orally on days 1, 7, and 13 to measure total drug exposure was analyzed by the linear up/log down trapezoidal rule using noncompartmental methods with Phoenix WinNonlin® (version 8.0; Pharsight Corporation, Mountain View, CA).
Time Frame: 0 to 24 hours postdose on days 1, 7, and 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*ng/ml
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 12
hr*ng/ml
  Day 1 (phase 1) | 991.25 (378.02)
  Day 7 (phase 2) | 1929.78 (631.58)
  Day 13 (phase 3) | 1939 (748.78)

3. Primary Outcome: Maximum Total Plasma Concentration (Cmax) for Rivaroxaban
Description: Maximum total plasma concentration (Cmax) following a single dose of rivaroxaban 10 mg orally on days 1, 7, and 13 was analyzed using noncompartmental methods with Phoenix WinNonlin® (version 8.0; Pharsight Corporation, Mountain View, CA). Cmax for rivaroxaban was obtained directly by visual inspection of the plasma concentration versus time over 24 hours postdose.
Time Frame: Up to 24 hours postdose on days 1, 7, and 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 12
ng/mL
  Day 1 (phase 1) | 128.6 (42.39)
  Day 7 (phase 2) | 192.25 (61.72)
  Day 13 (phase 3) | 196.17 (62.27)

4. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) for Rivaroxaban
Description: Time to maximum plasma concentration for Rivaroxaban following a single dose of rivaroxaban 10 mg orally on days 1, 7, and 13 was analyzed using noncompartmental methods with Phoenix WinNonlin® (version 8.0; Pharsight Corporation, Mountain View, CA). Tmax for rivaroxaban was obtained directly by visual inspection of the plasma concentration versus time over 24 hours postdose.
Time Frame: Up to 24 hours postdose on days 1, 7, and 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 12
Hours
  Day 1 (phase 1) | 2.5 (1.38)
  Day 7 (phase 2) | 4.1 (1.26)
  Day 13 (phase 3) | 3.02 (1.29)

5. Primary Outcome: Terminal Elimination Half-life (t½) for Rivaroxaban
Description: Terminal elimination half-life (t½) for Rivaroxaban following a single dose of rivaroxaban 10 mg orally on days 1, 7, and 13 was analyzed using noncompartmental methods with Phoenix WinNonlin® (version 8.0; Pharsight Corporation, Mountain View, CA). The apparent elimination rate constant (λZ) was determined by calculating the absolute value of the slope of the log-linear regression of at least 3 points of the plasma concentration-time plot. The t½ was calculated as 0.693/apparent elimination rate constant (λZ).
Time Frame: Up to 24 hours postdose on days 1, 7, and 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 12
Hours
  Day 1 (phase 1) | 5.65 (0.84)
  Day 7 (phase 2) | 8.19 (2.52)
  Day 13 (phase 3) | 7.49 (1.68)

6. Primary Outcome: Apparent Oral Clearance (CL/F) for Rivaroxaban
Description: Apparent oral clearance (CL/F) for Rivaroxaban following a single dose of rivaroxaban 10 mg orally on days 1, 7, and 13 was analyzed using noncompartmental methods with Phoenix WinNonlin® (version 8.0; Pharsight Corporation, Mountain View, CA). CL/F was calculated as 10 mg ÷ AUC0-tau for rivaroxaban.
Time Frame: Up to 24 hours postdose on days 1, 7, and 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 12
L/hr
  Day 1 (phase 1) | 11.04 (4.69)
  Day 7 (phase 2) | 4.92 (1.77)
  Day 13 (phase 3) | 5.19 (2.11)

7. Primary Outcome: Apparent Volume of Distribution (V/F) for Rivaroxaban
Description: Apparent volume of distribution (V/F) for Rivaroxaban following a single dose of rivaroxaban 10 mg orally on days 1, 7, and 13 was analyzed using noncompartmental methods with Phoenix WinNonlin® (version 8.0; Pharsight Corporation, Mountain View, CA).
Time Frame: Up to 24 hours postdose on days 1, 7, and 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 12
Liter
  Day 1 (phase 1) | 89.94 (42.32)
  Day 7 (phase 2) | 56.22 (23.07)
  Day 13 (phase 3) | 52.84 (16.32)

8. Primary Outcome: Minimum Total Plasma Concentration (Cmin) for Rivaroxaban
Description: Minimum total plasma concentration (Cmin) for Rivaroxaban following a single dose of rivaroxaban 10 mg orally on days 1, 7, and 13 was analyzed using noncompartmental methods with Phoenix WinNonlin® (version 8.0; Pharsight Corporation, Mountain View, CA). Cmin for rivaroxaban was obtained directly by visual inspection of the plasma concentration versus times over 24 hours postdose.
Time Frame: Up to 24 hours postdose on days 1, 7, and 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
Number analyzed (Participants) | 12
ng/mL
  Day 1 (phase 1) | 6.93 (3.43)
  Day 7 (phase 2) | 27.32 (13.25)
  Day 13 (phase 3) | 24.43 (14.38)

ADVERSE EVENTS:
Time Frame: 23 days
Arm/Group | Pharmacokinetic Study in Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 8/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pharmacokinetic Study in Healthy Volunteers (N=12)
Dizziness (Cardiac disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Blood bicarbonate decreased (Investigations) | 5
Blood bilirubin increased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Glomerular filtration rate decreased (Investigations) | 2
Haemoglobin decreased (Investigations) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/06/NCT03864406/Prot_SAP_000.pdf